CLINICAL TRIAL: NCT06393374
Title: A Phase 3, Randomized, Open-label, Study to Compare the Efficacy and Safety of Adjuvant MK-2870 in Combination With Pembrolizumab (MK-3475) Versus Treatment of Physician's Choice (TPC) in Participants With Triple-Negative Breast Cancer (TNBC) Who Received Neoadjuvant Therapy and Did Not Achieve a Pathological Complete Response (pCR) at Surgery
Brief Title: Sacituzumab Tirumotecan (MK-2870) Plus Pembrolizumab Versus TPC in TNBC Who Did Not Achieve pCR (MK-2870-012)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2870-012; 2023-504962-52-00 (Registry Identifier: EU CT); U1111-1289-8264 (Registry Identifier: UTN); jRCT2031240476 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — pembrolizumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + sacituzumab tirumotecan (Experimental): Participants receive pembrolizumab every 6 weeks (q6w) in combination with sacituzumab tirumotecan every 2 weeks (q2w) for 24 weeks. In addition, participants receive an antihistamine, an H2 antagonist of investigator's choice, acetaminophen (or equivalent), and dexamethasone (or equivalent) per each drug's product label prior to sacituzumab tirumotecan infusions.
  Interventions: Biological: Pembrolizumab; Biological: Sacituzumab tirumotecan
- Treatment of Physician's Choice (Active Comparator): Participants receive pembrolizumab q6w or pembrolizumab q6w in combination with capecitabine (twice daily [BID] on Days 1 to 14 and 22 to 35 every 42 days x 4 [2 weeks 1, 1 week off]) for 24 weeks.
  Interventions: Biological: Pembrolizumab; Drug: Capecitabine

INTERVENTIONS:
Biological: Pembrolizumab — Pembrolizumab 400 mg intravenous (IV) infusion q6w
  Other Names: KEYTRUDA®; MK-3475; SCH 900475
Biological: Sacituzumab tirumotecan — Sacituzumab tirumotecan 4 mg/kg IV infusion q2w
  Other Names: MK-2870
  Arms: Pembrolizumab + sacituzumab tirumotecan
Drug: Capecitabine — Capecitabine 1000 mg/m^2 to 1250 mg/m^2 by mouth BID
  Other Names: XELODA
  Arms: Treatment of Physician's Choice

SUMMARY:
This is a randomized, open-label study comparing the efficacy and safety of adjuvant sacituzumab tirumotecan (MK-2870) in combination with pembrolizumab compared to treatment of physician's choice (TPC) in participants with triple-negative breast cancer (TNBC) who received neoadjuvant therapy and did not achieve a pathological complete response (pCR) at surgery. The primary objective is to compare sacituzumab tirumotecan plus pembrolizumab to TPC (pembrolizumab or pembrolizumab plus capecitabine) with respect to invasive disease-free survival (iDFS) per investigator assessment. It is hypothesized that sacituzumab tirumotecan plus pembrolizumab is superior to TPC with respect to iDFS per investigator assessment.

ELIGIBILITY:
Inclusion Criteria:

* Has centrally confirmed TNBC, as defined by the most recent American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines
* Has no evidence of locoregional or distant relapse, as assessed by the treating physician
* Had neoadjuvant treatment based on the KEYNOTE-522 regimen (pembrolizumab with carboplatin/taxanes and pembrolizumab with anthracycline-based chemotherapy) followed by surgery according to National Comprehensive Cancer Network (NCCN) treatment guidelines for TNBC
* Had adequate excision and surgical removal of all clinically evident disease in the breast and/or lymph nodes and have adequately recovered from surgery
* Has non-pathologic complete response at surgery
* Is able to continue on adjuvant pembrolizumab
* Randomization must be conducted within 16 weeks from surgical resection
* Completed adjuvant radiation therapy (if indicated) and recovered before randomization
* Has provided tissue from the surgical resection for central laboratory determination of trophoblast cell surface antigen 2 (TROP2) status
* If capable of producing sperm, the participant agrees to the following during the intervention period and for at least the time needed to eliminate each study intervention after the last dose of study intervention (120 days for sacituzumab tirumotecan and 95 days for capecitabine [no restriction for pembrolizumab]): agrees to refrain from donating sperm AND is either abstinent and agrees to remain abstinent or uses highly effective contraception
* For females (assigned at birth), is not pregnant or breastfeeding and ≥1 of the following applies: is not a participant of childbearing potential (POCBP) OR is a POCBP and uses highly effective contraception after the last dose of study intervention (210 days for sacituzumab tirumotecan, 120 days for pembrolizumab, and 185 days for capecitabine). Abstains from breastfeeding during the study intervention period and for at least 120 days after study intervention
* Participants who have AEs due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline (except alopecia)
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy (ART)
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 assessed within 7 days before first dose of study treatment
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B birus (HBV) antiviral therapy for at least 4 weeks, and have undetectable HBV viral load prior to randomization

Exclusion Criteria:

* Has a known germline breast cancer gene (BRCA) mutation (deleterious or suspected deleterious) and is eligible for adjuvant therapy with olaparib where olaparib is approved and available
* Has Grade >2 peripheral neuropathy
* History of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis, or chronic diarrhea)
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, uncontrolled symptomatic arrhythmia, prolongation of QTcF interval to >480 ms, and/or other serious cardiovascular and cerebrovascular diseases within 6 months prior to study intervention
* Received prior treatment with a trophoblast cell-surface antigen 2 (TROP2)-directed antibody drug conjugate (ADC) or a topoisomerase I inhibitor-containing ADC
* Received anticancer therapy in the adjuvant phase including but not limited to chemotherapy, small molecule anticancer drugs, poly (adenosine diphosphate ribose) polymerase (PARP) inhibitors, ADCs, and/or immunotherapy, with the exception of adjuvant radiation therapy
* Is currently receiving a strong inducer/inhibitor of cytochrome P450 3A4 (CYP3A4) that cannot be discontinued for the duration of the study. The required washout period before starting sacituzumab tirumotecan is 2 weeks
* Except for pembrolizumab as neoadjuvant therapy for early-stage TNBC: received prior therapy with an anti-programmed cell death 1 protein (anti-PD-1), anti-programmed cell death ligand 1 (anti-PD-L1), or anti-PD-L2 agent, or with an agent directed to another stimulatory or coinhibitory T-cell receptor (eg, cytotoxic T-lymphocyte-associated protein-4 [CTLA-4], OX-40 [cluster of differentiation (CD) 134], or CD137)
* Except for chemotherapy as neoadjuvant therapy for early-stage TNBC: Received prior systemic anticancer therapy including investigational agents within 4 weeks before randomization
* Received prior radiotherapy within 3 weeks of start of study intervention or required corticosteroids for radiation related toxicities that cannot be discontinued before the first dose of study intervention
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines are allowed
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* Has known additional malignancy that is progressing or has required active treatment within the past 5 years
* Has diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study medication
* Has active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid) is allowed
* Has history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has active infection requiring systemic therapy
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has concurrent active hepatitis B and hepatitis C virus infection
* Has history of allogeneic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1530 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2030-12-16 (Estimated); Study Completion 2037-12-14 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-Free Survival (iDFS) | Up to ~77 months
  iDFS is the time from randomization to invasive local, regional, or distant recurrence, invasive contralateral breast cancer, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to ~101 months
  OS is the time from randomization to death due to any cause.
Distant recurrence-free survival (DRFS) | Up to ~101 months
  DRFS is the time from randomization to distant recurrence or death due to any cause, whichever occurs first.
Change from baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Global Health Status (Item 29) and Quality of Life (Item 30) Combined Score | Baseline and up to ~60 months
  EORTC QLQ-C30 is a 30-item scale to assess the overall quality of life in cancer patients. The overall functioning score is based on participant responses that are scored on a 7-point scale (1 = "Very poor" to 7 = "Excellent"). Higher scores indicate better overall health status.
Change from baseline in EORTC QLQ-C30 Physical Functioning (Items 1-5) Combined Score | Baseline and up to ~60 months
  EORTC QLQ-C30 is a 30-item scale to assess the overall quality of life of cancer patients. The physical functioning score is based on participant responses to questions that scored on a 4-point scale (1 = 'Not at All' to 4 = 'Very Much'). Higher scores indicate better physical functioning.
Change from baseline in EORTC QLQ-C30 Role Functioning (Items 6 and 7) Combined Score | Baseline and up to ~60 months
  EORTC QLQ-C30 is a 30-item scale to assess the overall quality of life of cancer patients. The role functioning score is based on participant responses to questions that scored on a 4-point scale (1 = 'Not at All' to 4 = 'Very Much'). Higher scores indicate better role functioning.
Change from baseline in EORTC QLQ-C30 Fatigue (Items 10, 12, and 18) Combined Score | Baseline and up to ~60 months
  EORTC QLQ-C30 is a 30-item scale to assess the overall quality of life of cancer patients. Participant responses to questions about their fatigue are scored on a 4-point scale (1 = "Not at All" to 4 = "Very Much"). Lower scores indicate a better level of fatigue.
Number of participants who experience one or more adverse events (AEs) | Up to ~42 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants who discontinue study intervention due to an AE | Up to 24 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (275):
- United States (73):
  - Infirmary Cancer Care ( Site 0001), Mobile, Alabama
  - Ironwood Cancer & Research Centers-Research ( Site 0054), Chandler, Arizona
  - MemorialCare Orange Coast Medical Center ( Site 9501), Fountain Valley, California
  - Scripps Cancer Center ( Site 0052), La Jolla, California
  - Cancer and Blood Specialty Clinic ( Site 0008), Los Alamitos, California
  - Kaiser Permanente - Oakland ( Site 0079), Oakland, California
  - Profound Research LLC ( Site 0105), Oceanside, California
  - Kaiser Permanente - Roseville ( Site 0081), Roseville, California
  - Kaiser Permanente - San Francisco ( Site 0080), San Francisco, California
  - Kaiser Permanente - Santa Clara ( Site 0082), Santa Clara, California
  - Kaiser Permanente Vallejo Medical Center ( Site 0060), Vallejo, California
  - Kaiser Permanente - Walnut Creek ( Site 0078), Walnut Creek, California
  - Bass Medical Group ( Site 0089), Walnut Creek, California
  - Cancer Centers of Colorado St. Mary's Regional Hospital ( Site 0046), Grand Junction, Colorado
  - Yale Cancer Center ( Site 0053), New Haven, Connecticut
  - Comprehensive Hematology Oncology ( Site 0091), St. Petersburg, Florida
  - Cleveland Clinic Martin North Hospital ( Site 0114), Stuart, Florida
  - Archbold Memorial Hospital-Lewis Hall Singletary Oncology Center ( Site 0040), Thomasville, Georgia
  - Illinois Cancer Specialists (ICS) ( Site 8010), Arlington Heights, Illinois
  - Orchard Healthcare Research Inc. ( Site 0014), Skokie, Illinois
  - Northwest Cancer Center - Dyer Clinic ( Site 0097), Dyer, Indiana
  - Parkview Research Center at Parkview Regional Medical Center ( Site 0011), Fort Wayne, Indiana
  - Cancer Center of Kansas ( Site 0004), Wichita, Kansas
  - Saint Elizabeth Medical Center Edgewood-Cancer Care Center ( Site 0044), Edgewood, Kentucky
  - CHRISTUS St. Frances Cabrini Hospital Center for Cancer Care ( Site 0109), Alexandria, Louisiana
  - Ochsner LSU Health - Monroe Medical Center, Family Medicine Clinic ( Site 0063), Monroe, Louisiana
  - Louisiana State University Health Sciences Shreveport ( Site 0029), Shreveport, Louisiana
  - Holy Cross Hospital ( Site 0069), Silver Spring, Maryland
  - Profound Research LLC ( Site 0074), Royal Oak, Michigan
  - The University of Mississippi Medical Center-Cancer Center and Research Institute ( Site 0043), Jackson, Mississippi
  - SSM Health Cancer Care - Fenton ( Site 0088), Fenton, Missouri
  - Lake Regional Hospital ( Site 0009), Osage Beach, Missouri
  - Siteman Cancer Center ( Site 0099), St Louis, Missouri
  - New Mexico Oncology Hematology Consultants Ltd. ( Site 0090), Albuquerque, New Mexico
  - CHRISTUS St. Vincent Regional Cancer Center ( Site 0118), Santa Fe, New Mexico
  - Memorial Sloan Kettering Cancer Center ( Site 0067), New York, New York
  - Clinical Research Alliance ( Site 0086), Westbury, New York
  - Levine Cancer Institute ( Site 0083), Charlotte, North Carolina
  - Sanford Cancer Center Bismarck ( Site 0058), Bismarck, North Dakota
  - Sanford Fargo Medical Center-Roger Maris Cancer Center ( Site 0056), Fargo, North Dakota
  - Altru Cancer Center ( Site 0104), Grand Forks, North Dakota
  - Cleveland Clinic - Mercy Hospital ( Site 0057), Canton, Ohio
  - Tri-County Hematology & Oncology Associates, Inc. ( Site 0076), Massillon, Ohio
  - Genesis Healthcare System ( Site 0025), Zanesville, Ohio
  - Hightower Clinical, LLC ( Site 0085), Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute, LLC ( Site 0041), Tulsa, Oklahoma
  - Providence Portland Medical Center ( Site 0116), Portland, Oregon
  - Providence Oncology and Hematology Care Clinic - Westside ( Site 0126), Portland, Oregon
  - Sidney Kimmel Cancer Center at Jefferson ( Site 0049), Philadelphia, Pennsylvania
  - Sanford Cancer Center ( Site 0059), Sioux Falls, South Dakota
  - West Cancer Center and Research Institute ( Site 0084), Germantown, Tennessee
  - Baptist Cancer Center ( Site 0101), Memphis, Tennessee
  - One Oncology - Tennessee Oncology ( Site 0098), Nashville, Tennessee
  - SCRI Oncology Partners ( Site 7000), Nashville, Tennessee
  - Tennessee Oncology ( Site 0111), Nashville, Tennessee
  - Nashville General Hospital ( Site 0072), Nashville, Tennessee
  - Vanderbilt Health One Hundred Oaks ( Site 0042), Nashville, Tennessee
  - Harrington Cancer Center ( Site 0061), Amarillo, Texas
  - Texas Oncology - DFW ( Site 8000), Dallas, Texas
  - Parkland Health & Hospital System ( Site 0096), Dallas, Texas
  - University of Texas Southwestern Medical Center ( Site 0032), Dallas, Texas
  - Texas Oncology - Northeast Texas ( Site 8005), Flower Mound, Texas
  - John Peter Smith Hospital ( Site 0106), Fort Worth, Texas
  - Oncology Consultants P.A. ( Site 0107), Houston, Texas
  - Doctors Hospital of Laredo ( Site 0068), Laredo, Texas
  - The University of Texas Health Science Center at Tyler dba UT Health East Texas HOPE Cancer Center ( Site 0055), Tyler, Texas
  - Texas Oncology - Gulf Coast ( Site 8009), Webster, Texas
  - Intermountain Medical Center ( Site 0113), Murray, Utah
  - Hematology Oncology Associates of Fredericksburg ( Site 9550), Fredericksburg, Virginia
  - Bon Secours Memorial Regional Medical Center-Oncology Research Department ( Site 0020), Midlothian, Virginia
  - Virginia Cancer Institute ( Site 0034), Richmond, Virginia
  - Northwest Medical Specialties, PLLC ( Site 0093), Tacoma, Washington
  - SSM Health Dean Medical Group ( Site 0087), Madison, Wisconsin
- Argentina (7):
  - Hospital Aleman-Oncology ( Site 0501), Capital Federal, Buenos Aires
  - Hospital Británico de Buenos Aires-Oncology ( Site 0502), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto de Oncología Angel H. Roffo ( Site 0503), Buenos Aires, Buenos Aires F.D.
  - Instituto Alexander Fleming-Alexander Fleming ( Site 0509), Buenos Aires, Buenos Aires F.D.
  - Sanatorio Parque ( Site 0512), Rosario, Santa Fe Province
  - Sanatorio Finochietto ( Site 0513), Buenos Aires
  - Centro de Educación Médica e Investigaciones clínicas "Dr. Norberto Quirno" (CEMIC) ( Site 0508), Buenos Aires
- Australia (4):
  - Macquarie University-MQ Health Clinical Trials Unit ( Site 2703), Macquarie University, New South Wales
  - Westmead Hospital ( Site 2700), Westmead, New South Wales
  - Royal Brisbane and Women's Hospital-Medical Oncology Clinical Trials Unit, Cancer Care Services ( Site 2701), Brisbane, Queensland
  - Frankston Hospital-Oncology and Haematology ( Site 2704), Frankston, Victoria
- Austria (5):
  - Medizinische Universitaet Innsbruck ( Site 1200), Innsbruck, Tyrol
  - Kepler Universitätsklinikum-Department for Oncology and Hematology ( Site 1206), Linz, Upper Austria
  - Klinikum Wels-Grieskirchen ( Site 1205), Wels, Upper Austria
  - Uniklinikum Salzburg-Universitätsklinik für Innere Medizin III der PMU mit Hämatologie, internistis ( Site 1202), Salzburg
  - Medizinische Universität Wien-Universitätsklinik für Innere Medizin I, Klinische Abteilung für Onko ( Site 1201), Vienna
- Belgium (3):
  - Cliniques universitaires Saint-Luc-Medical Oncology ( Site 0901), Brussels, Bruxelles-Capitale, Region de
  - AZ Maria Middelares-IKG ( Site 0903), Ghent, Oost-Vlaanderen
  - Université Catholique de Louvain-Namur - Centre Hospitalier -Oncology ( Site 0902), Namur
- Brazil (6):
  - PRONUTRIR-CLINICAL RESEARCH ( Site 0609), Fortaleza, Ceará
  - Oncoclínica Oncologistas Associados-Clinical Research ( Site 0607), Teresina, Piauí
  - Hospital do Câncer Mãe de Deus ( Site 0604), Porto Alegre, Rio Grande do Sul
  - Instituto de Oncologia Saint Gallen ( Site 0614), Santa Cruz do Sul, Rio Grande do Sul
  - Instituto do Câncer Brasil - Unidade Taubaté ( Site 0608), Taubaté, São Paulo
  - IBCC - Núcleo de Pesquisa e Ensino ( Site 0601), São Paulo
- Canada (15):
  - Cross Cancer Institute ( Site 0407), Edmonton, Alberta
  - BC Cancer Vancouver ( Site 0404), Vancouver, British Columbia
  - CancerCare Manitoba ( Site 0411), Winnipeg, Manitoba
  - The Moncton Hospital ( Site 0401), Moncton, New Brunswick
  - QEII Health Sciences Centre - Victoria General Site ( Site 0418), Halifax, Nova Scotia
  - Southlake Health ( Site 0413), Newmarket, Ontario
  - The Ottawa Hospital - General Campus ( Site 0414), Ottawa, Ontario
  - North York General Hospital ( Site 0415), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0400), Toronto, Ontario
  - Centre Intégré de Santé et de Services Sociaux de la Montérégie-Centre ( Site 0417), Greenfield Park, Quebec
  - CIUSSS de l'Est-de-l'Île-de-Montréal ( Site 0419), Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal ( Site 0403), Montreal, Quebec
  - Jewish General Hospital ( Site 0416), Montreal, Quebec
  - Centre intégré de santé et de services sociaux du Bas Saint-Laurent- Hôpital régional de Rimouski ( Site 0409), Rimouski, Quebec
  - Centre integre universitaire de sante et de services sociaux de la Mauricie-et-du-centre-du-quebec ( Site 0406), Trois-Rivières, Quebec
- Colombia (4):
  - Clinica Somer ( Site 3704), Rionegro, Antioquia
  - FUNDACION CTIC CENTRO DE TRATAMIENTO E INVESTIGACION SOBRE CANCER LUIS CARLOS SARMIENTO ANGULO ( Site 3700), Bogotá, Bogota D.C.
  - Instituto Nacional De Cancerologia ( Site 3701), Bogotá, Bogota D.C.
  - Sociedad de Oncología Y Hematología del Cesar S.A.S. ( Site 3705), Valledupar, Cesar Department
- Czechia (6):
  - Masarykuv onkologicky ustav-Klinika komplexni onkologicke pece ( Site 1005), Brno, Brno-mesto
  - Nemocnice Ceske Budejovice-Onkologicke oddeleni ( Site 1007), České Budějovice, Jihočeský kraj
  - Fakultni nemocnice Olomouc-Onkologicka klinika ( Site 1006), Olomouc, Olomoucký kraj
  - Vseobecna fakultni nemocnice v Praze-Onkologická klinika VFN ( Site 1002), Prague, Praha 2
  - Fakultni Thomayerova nemocnice - Onkologicka klinika 1. LF UK a FTN ( Site 1008), Prague, Praha 4
  - Fakultni nemocnice v Motole-Onkologicka klinika 2. LF UK a FN Motol ( Site 1000), Prague, Praha 5
- Denmark (3):
  - Herlev og Gentofte Hospital. ( Site 3203), Herlev, Capital Region
  - Odense Universitetshospital ( Site 3201), Odense C, Region Syddanmark
  - Sygehus Soenderjylland ( Site 3204), Sønderborg, Region Syddanmark
- Finland (3):
  - Tampereen yliopistollinen sairaala ( Site 1102), Tampere, Pirkanmaa
  - Turku University Hospital-Department of Oncology ( Site 1103), Turku, Southwest Finland
  - Helsinki University Hospital - Comprehensive Cancer Center (HYKS - Syöpäkeskus) ( Site 1100), Helsinki, Uusimaa
- France (18):
  - Centre Antoine-Lacassagne ( Site 1308), Nice, Alpes-Maritimes
  - Centre Hospitalier de la Côte Basque ( Site 1315), Bayonne, Aquitaine
  - CENTRE LEON BERARD ( Site 1300), Lyon Cedex08, Auvergne-Rhône-Alpes
  - Centre Jean Perrin - Centre Régional de Lutte contre le Cancer d'Auvergne ( Site 1307), Clermont-Ferrand, Auvergne
  - Institut Paoli-Calmettes ( Site 1309), Marseille, Bouches-du-Rhone
  - Centre François Baclesse ( Site 1318), Caen, Calvados
  - Centre Georges François Leclerc ( Site 1312), Dijon, Cote-d Or
  - CHU Besançon ( Site 1311), Besançon, Doubs
  - Hôpital Privé Drôme-Ardèche ( Site 1301), Valence, Drome
  - CHRU Brest - Hopital Cavale Blanche ( Site 1304), Brest, Finistere
  - Clinique Tivoli Ducos ( Site 1322), Bordeaux, Gironde
  - Hôpital Franco-Britannique - Fondation Cognacq-Jay ( Site 1321), Levallois-Perret, Hauts-de-Seine
  - Institut de Cancérologie de l'Ouest ( Site 1305), Saint-Herblain, Loire-Atlantique
  - Institut de Cancérologie de l'Ouest ( Site 1316), Angers, Maine-et-Loire
  - Centre de Cancerologie Les Dentellieres ( Site 1306), Valenciennes, Nord
  - Centre Hospitalier de Pau ( Site 1302), Pau, Pyrenees-Atlantiques
  - Centre Henri Becquerel ( Site 1319), Rouen, Seine-Maritime
  - Hôpital Tenon ( Site 1303), Paris
- Germany (13):
  - Klinikum Ludwigsburg-Klinik für Geburtshilfe und Frauenheilkunde ( Site 1405), Ludwigsburg, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen-Frauenklinik ( Site 1415), Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen-Klinik für Gynäkologie und Geburtshilfe ( Site 1400), Erlangen, Bavaria
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen-Frauenklinik Brustzentrum ( Site 1402), Munich, Bavaria
  - Klinikum Ernst von Bergmann-Frauenklinik ( Site 1408), Potsdam, Brandenburg
  - Franziskus-Hospital Harderberg ( Site 1404), Georgsmarienhütte, Lower Saxony
  - Universitaetsklinikum Duesseldorf-Klinik für Frauenheilkunde & Geburtshilfe ( Site 1409), Düsseldorf, North Rhine-Westphalia
  - Kliniken Essen-Mitte, Evangelische Huyssens-Stiftung-Klinik für Senologie/ Brustzentrum ( Site 1401), Essen, North Rhine-Westphalia
  - Evangelisches Krankenhaus Bethesda Mönchengladbach-Brustzentrum Niederrhein ( Site 1406), Mönchengladbach, North Rhine-Westphalia
  - Universitätsmedizin Johannes Gutenberg Universität Mainz-Klinik und Poliklinik für Geburtshilfe und ( Site 1418), Mainz, Rhineland-Palatinate
  - CaritasKlinikum Saarbruecken St. Theresia ( Site 1410), Saarbrücken, Saarland
  - Universitätsklinikum Schleswig-Holstein ( Site 1411), Lübeck, Schleswig-Holstein
  - Helios Klinikum Berlin-Buch-Klinik für Gynäkologie und Geburtshilfe ( Site 1413), Berlin
- Greece (6):
  - UNIVERSITY HOSPITAL OF PATRAS-DIVISION OF ONCOLOGY ( Site 1509), Pátrai, Achaia
  - Errikos Dunant Hospital Center-1st Medical Oncology Dept. ( Site 1508), Athens, Attica
  - Aretaieio Hospital Oncology Unit ( Site 1505), Athens, Attica
  - University General Hospital of Larissa ( Site 1503), Larissa, Thessaly
  - European Interbalkan Medical Center ( Site 1502), Thessaloniki
  - European Interbalkan Medical Center ( Site 1507), Thessaloniki
- Hong Kong (2):
  - Queen Mary Hospital ( Site 3600), Hong Kong
  - Hong Kong United Oncology Centre ( Site 3601), Kowloon
- Ireland (3):
  - Bon Secours Cork Hospital ( Site 1600), Cork
  - St. Vincent's University Hospital-Medical Oncology Research Department ( Site 1601), Dublin
  - University College Hospital - Galway ( Site 1602), Galway
- Israel (5):
  - Soroka Medical Center-Oncology ( Site 1704), Beersheba
  - Hadassah Medical Center ( Site 1700), Jerusalem
  - Rabin Medical Center ( Site 1702), Petah Tikva
  - Sheba Medical Center-ONCOLOGY ( Site 1701), Ramat Gan
  - Sourasky Medical Center ( Site 1705), Tel Aviv
- Italy (14):
  - University of Naples Federico II-Dipartimento di Medicina Clinica e Chirurgia ( Site 1803), Naples, Campania
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale-S.C. Oncologia Clinica Sperimentale di Senologia ( Site 1800), Napoli, Campania
  - Humanitas Istituto Clinico Catanese ( Site 1811), Misterbianco, Catania
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori" ( Site 1807), Meldola (FC), Forli-Cesena
  - CRO-IRCCS ( Site 1808), Aviano, Friuli Venezia Giulia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS -Medical Oncology ( Site 1802), Rome, Lazio
  - Azienda Ospedaliera Spedali Civili di Brescia ( Site 1812), Brescia, Lombardy
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 1801), Milan, Lombardy
  - Istituto Europeo di Oncologia IRCCS-Divisione di Senologia Medica ( Site 1809), Milan, Lombardy
  - Fondazione IRCCS San Gerardo dei Tintori ( Site 1813), Monza, Lombardy
  - Azienda Ospedaliera Universitaria Careggi ( Site 1805), Florence, Tuscany
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola ( Site 1810), Bologna
  - Ospedale San Raffaele-Oncologia Medica ( Site 1814), Milan
  - Azienda Ospedaliero Universitaria Maggiore della Carità-SCDU ONCOLOGIA ( Site 1804), Novara
- Japan (24):
  - Nagoya City University Hospital ( Site 3414), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 3403), Kashiwa, Chiba
  - Hokkaido University Hospital ( Site 3400), Sapporo, Hokkaido
  - Tokai University Hospital ( Site 3413), Isehara, Kanagawa
  - St. Marianna University Hospital ( Site 3405), Kawasaki, Kanagawa
  - Kitasato University Hospital ( Site 3411), Sagamihara, Kanagawa
  - Kanagawa Cancer Center ( Site 3412), Yokohama, Kanagawa
  - Mie University Hospital ( Site 3423), Tsu, Mie-ken
  - Tohoku University Hospital ( Site 3422), Sendai, Miyagi
  - The University of Osaka Hospital ( Site 3416), Suita, Osaka
  - Saitama Medical University International Medical Center ( Site 3402), Hidaka, Saitama
  - Juntendo University Hospital ( Site 3408), Bunkyo, Tokyo
  - Cancer Institute Hospital of JFCR ( Site 3404), Koto, Tokyo
  - Showa Medical University Hospital ( Site 3406), Shinagawa, Tokyo
  - Tokyo Medical University Hospital ( Site 3407), Shinjuku, Tokyo
  - National Center for Global Health and Medicine ( Site 3409), Shinjuku, Tokyo
  - Fukushima Medical University Hospital ( Site 3401), Fukushima
  - Gifu University Hospital ( Site 3426), Gifu
  - Hiroshima City Hiroshima Citizens Hospital ( Site 3418), Hiroshima
  - Social medical corporation Hakuaikai Sagara Hospital ( Site 3421), Kagoshima
  - Kumamoto University Hospital ( Site 3420), Kumamoto
  - Kyoto University Hospital ( Site 3415), Kyoto
  - Okayama University Hospital ( Site 3425), Okayama
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute ( Site 3417), Osaka
- Malaysia (2):
  - Prince Court Medical Centre ( Site 2802), Kuala Lumpur
  - Pantai Hospital Kuala Lumpur ( Site 2801), Kuala Lumpur
- Mexico (6):
  - CENEIT Oncologicos ( Site 0706), Mexico City, Mexico City
  - Grupo Médico ASSET ( Site 0705), Mexico City, Mexico City
  - Health Pharma Professional Research S.A. de C.V: ( Site 0709), Mexico City, Mexico City
  - COI Centro Oncologico Internacional S.A.P.I. de C.V. ( Site 0712), Mexico City, Mexico City
  - Oncare - Unidad Valle ( Site 0713), San Pedro Garza García, Nuevo León
  - CENTRO MEDICO ZAMBRANO HELLION ( Site 0711), San Pedro Garza García, Nuevo León
- Norway (3):
  - Drammen Sykehus, Vestre Viken HF ( Site 2001), Drammen, Buskerud
  - Stavanger Universitetssykehus ( Site 2004), Stavanger, Rogaland
  - Oslo universitetssykehus, Radiumhospitalet ( Site 2002), Oslo
- Poland (9):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 2102), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Oddzial w Krakowie ( Site 2120), Krakow, Lesser Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworów Piersi i Chirurgii ( Site 2100), Warsaw, Masovian Voivodeship
  - Mazowiecki Szpital Onkologiczny-BREAST CANCER ( Site 2101), Wieliszew, Masovian Voivodeship
  - Bialostockie Centrum Onkologii ( Site 2105), Bialystok, Podlaskie Voivodeship
  - Szpitale Pomorskie Sp. z o. o.-Oddział Onkologii Klinicznej ( Site 2113), Gdynia, Pomeranian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach-Centrum Diagnostyki i Leczenia Chorob Piersi ( Site 2110), Gliwice, Silesian Voivodeship
  - Zachodniopomorskie Centrum Onkologii ( Site 2108), Szczecin, West Pomeranian Voivodeship
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zakl-Klinika Onkologii Klinicznej, Dzial Ch ( Site 2118), Kielce, Świętokrzyskie Voivodeship
- Portugal (4):
  - Unidade Local de Saude Amadora/Sintra - Hospital Prof Dr Fernando Fonseca ( Site 2203), Amadora, Lisbon District
  - Fundacao Champalimaud ( Site 2200), Lisbon
  - Unidade Local de Saude de Santa Maria - Hospital de Santa Maria ( Site 2201), Lisbon
  - Instituto Portugues de Oncologia do Porto ( Site 2202), Porto
- National Cancer Centre Singapore-Medical Oncology ( Site 3002), Singapore, Central Singapore, Singapore
- South Korea (5):
  - Seoul National University Hospital-Internal Medicine ( Site 3102), Seoul
  - Severance Hospital, Yonsei University Health System-Medical oncology ( Site 3100), Seoul
  - Asan Medical Center-Department of Oncology ( Site 3103), Seoul
  - Gangnam Severance Hospital, Yonsei University Health System-Medical Oncology, Internal Medicine ( Site 3104), Seoul
  - Samsung Medical Center-Division of Hematology/Oncology ( Site 3101), Seoul
- Spain (10):
  - HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO-Medical Oncology ( Site 2304), Seville, Andalusia
  - Institut Català d'Oncologia - L'Hospitalet-Medical Oncology ( Site 2305), L'Hospitalet de Llobregat, Barcelona
  - CHUAC-Hospital Teresa Herrera-MEDICAL ONCOLOGY ( Site 2307), A Coruña, La Coruna
  - Hospital Universitario Ramón y Cajal-Medical Oncology ( Site 2301), Madrid, Madrid, Comunidad de
  - HOSPITAL UNIVERSITARIO PUERTA DE HIERRO MAJADAHONDA-Medical Oncology ( Site 2308), Majadahonda, Madrid, Comunidad de
  - Fundación Instituto Valenciano de Oncología-Oncologico ( Site 2303), Valencia, Valenciana, Comunitat
  - Hospital Universitari Vall d'Hebron-Oncology ( Site 2300), Barcelona
  - Hospital Beata María Ana-oncology ( Site 2309), Madrid
  - Hospital Clinico San Carlos-Oncology Department ( Site 2306), Madrid
  - HOSPITAL CLINICO DE VALENCIA-Oncology ( Site 2302), Valencia
- Sweden (5):
  - Capio St. Gorans Sjukhus ( Site 3503), Stockholm, Stockholm County
  - Karolinska Universitetssjukhuset Solna ( Site 3500), Stockholm, Stockholm County
  - Akademiska Sjukhuset ( Site 3501), Uppsala, Uppsala County
  - Södra Älvsborg Sjukhus ( Site 3502), Borås, Västra Götaland County
  - Sahlgrenska Universitetssjukhuset. ( Site 3505), Gothenburg, Västra Götaland County
- Switzerland (5):
  - Spital Thun ( Site 2400), Thun, Canton of Bern
  - Clinique Générale-Beaulieu ( Site 2406), Geneva, Canton of Geneva
  - Brust-Zentrum ( Site 2401), Zurich, Canton of Zurich
  - Kantonsspital Graubünden-Medizin ( Site 2404), Chur, Kanton Graubünden
  - HFR Fribourg - Hôpital Cantonal ( Site 2402), Fribourg
- Turkey (Türkiye) (5):
  - Adana Medical Park Seyhan Hastanesi-Medikal Onkoloji ( Site 2501), Adana
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastırma Hastanesi-oncology ( Site 2504), Ankara
  - Memorial Ankara Hastanesi-Medical Oncology ( Site 2502), Ankara
  - Medipol Mega Universite Hastanesi-oncology ( Site 2503), Istanbul
  - Samsun Medical Park Hastanesi-medical oncology ( Site 2500), Samsun
- United Kingdom (6):
  - University Hospitals Bristol NHS Foundation Trust ( Site 2601), Bristol, Bristol, City of
  - The Royal Cornwall Hospital ( Site 2603), Truro, England
  - St Bartholomew's Hospital-Centre for Experimental Cancer Medicine ( Site 2602), London, London, City of
  - University College London Hospital ( Site 2604), London, London, City of
  - Western General Hospital ( Site 2607), Edinburgh, Midlothian
  - St James's University Hospital-Leeds Cancer Centre ( Site 2608), Leeds

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26291&tenant=MT_MSD_9011